CLINICAL TRIAL: NCT03673215
Title: A Phase Ia Dose-escalation Study to Access the Tolerability，Safety，Pharmacokinetics and Pharmacodynamics of Recombinant Human Thrombopoietin in the Patients With Different Degree of Liver Function Impairment
Brief Title: The Tolerability，Safety，PK/PD Study of rhTPO in the Patients With Liver Function Impairment
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3SBio-TPO-106
Record Dates: First submitted 2018-08-15; First posted 2018-09-17 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Thrombopoietin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- A (Experimental)
  Interventions: Drug: Recombinant human thrombopoietin
- B1 (Experimental)
  Interventions: Drug: Recombinant human thrombopoietin
- B2 (Placebo Comparator)
  Interventions: Drug: Placebo
- C1-1 (Experimental)
  Interventions: Drug: Recombinant human thrombopoietin
- C1-2 (Placebo Comparator)
  Interventions: Drug: Placebo
- C2-1 (Experimental)
  Interventions: Drug: recombinant human thrombopoietin
- C2-2 (Placebo Comparator)
  Interventions: Drug: placebo
- C3-1 (Experimental)
  Interventions: Drug: Recombinant human thrombopoietin
- C3-2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Recombinant human thrombopoietin — Recombinant human thrombopoietin will be administered single dose 300 U/Kg subcutaneous injection in the patients with liver function impairment classified as Child-Pugh class A
  Other Names: rhTPO
  Arms: A
Drug: Recombinant human thrombopoietin — Recombinant human thrombopoietin will be administered single dose 300 U/Kg subcutaneous injection in the patients with liver function impairment classified as Child-Pugh class B.
  Other Names: rhTPO
  Arms: B1
Drug: Placebo — Placebo will be administered single dose subcutaneous injection in the patients with liver function impairment classified as Child-Pugh class B.
  Arms: B2
Drug: Recombinant human thrombopoietin — Recombinant human thrombopoietin will be administered single dose 150 U/Kg subcutaneous injection in the patients with liver function impairment classified as Child-Pugh class C.
  Other Names: rhTPO
  Arms: C1-1
Drug: Placebo — Placebo will be administered single dose subcutaneous injection in the patients with liver function impairment classified as Child-Pugh class C
  Arms: C1-2
Drug: recombinant human thrombopoietin — Recombinant human thrombopoietin will be administered single dose 300 U/Kg subcutaneous injection in the patients with liver function impairment classified as Child-Pugh class C.
  Other Names: rhTPO
  Arms: C2-1
Drug: placebo — Placebo will be administered single dose subcutaneous injection in the patients with liver function impairment classified as Child-Pugh class C
  Arms: C2-2
Drug: Recombinant human thrombopoietin — Recombinant human thrombopoietin will be administered single dose 450 U/Kg subcutaneous injection in the patients with liver function impairment classified as Child-Pugh class C.
  Other Names: rhTPO
  Arms: C3-1
Drug: placebo — Placebo will be administered single dose subcutaneous injection in the patients with liver function impairment classified as Child-Pugh class C
  Arms: C3-2

SUMMARY:
The purpose of this study is to evaluate the tolerability, safety, pharmacokinetics and pharmacodynamics of recombinant human thrombopoietin in the patients with different degree of liver function impairment according Child- Pugh class.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, dose-escalation phase Ia study to evaluate the tolerability, safety, pharmacokinetics and pharmacodynamics of recombinant human thrombopoietin. According Child- Pugh class of liver function impairment and different dose of recombinant human thrombopoietin, nine arms be designed in this study. Each subject in Arm A will be only administered recombinant human thrombopoietin. Each subject in Arm B and C will be randomly assigned to accept either recombinant human thrombopoietin or placebo in 5:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with cirrhosis caused by chronic liver disease who have been diagnosed by biopsy/imaging (Child-Pugh class A, B, and C).
* 2. Life expectancy≥3 months.
* 3. Platelet count≤80×109/ L.
* 4. Fertile female subjects with a negative pregnancy test during the screening period and who agree to take effective contraceptive methods Throughout the study period will be eligible for this study.
* 5. Voluntary written informed consent.

Exclusion Criteria:

* 1 Subjects allergic to any component of investigational drug.
* 2 Subjects with cirrhosis caused by drug-induced liver injury.
* 3 Subjects with history of splenectomy or liver transplantation.
* 4 Liver cirrhosis with serious complications, including: hepatic encephalopathy, intractable ascites, upper gastrointestinal bleeding, etc.
* 5 Subjects with Liver failure.
* 6 Tthe presence of portal vein thrombosis or tumor thrombus was indicated by doppler ultrasound or CT or MRI and other imaging examinations within 3 months prior to the beginning of screening.
* 7 Subjects with history of arterial or venous thromboembolism, or with thromboembolic disease, or with high risk factors for thrombosis, or with a hereditary tendency to thrombosis, including Antithrombin III deficiency, etc.
* 8 Subjects with history of any disease other than chronic liver disease and cirrhosis that may result in decreased platelet count and/or abnormal platelet function, including aplastic anemia, myelodysplastic syndrome (MDS), bone marrow fibrosis, etc.;
* 9 Subjects with diseases with higher bleeding risk, such as coagulation factor deficiency or Vascular pseudohemophilia factor deficiency.
* 10 Subjects with severe infections that are not effectively controlled.
* 11 Past or present history with any serious disease except liver disease, including: angina, severe arrhythmia, myocardial infarction, heart failure, Cerebral hemorrhage, cerebral infarction, intracranial infection, Renal insufficiency( creatinine clearance rate ≤50 mL/min )，as well as any other diseases that have been judged by investigator to be unsuitable for this study.
* 12 Subjects who had undergone trans jugular intrahepatic portal shunt (TIPS);
* 13 Subjects with Anti-HIV positive antibodies or Anti- TPHA positive antibodies.
* 14 Subjects who received any therapy with increased platelet count within the 3 weeks or platelet transfusion within 2 weeks before randomization.
* 15 No more than 30 days or 5 half-lives after investigational drug treatment for other studies (whichever is longer).
* 16 Subjects with history of primary liver cancer, or an other malignant tumor.
* 17 patients with WHO≥grade 2 of existing active bleeding, or with history of active bleeding within 2 weeks before randomization.
* 18 Pregnant or breast-feeding women.
* 19 Women who have a pregnancy plan within 3 months.
* 20 Subjects with history of drug abuse and alcoholism within 6 months prior to enrollment.
* 21 Subjects who do not have the sufficient ability of understanding，communication and cooperation leading to failure to ensure compliance with protocol will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-10-08 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by the collection of adverse events | Up to 29 days
  To evaluate the adverse events (incidence, severity, outcome, causality with the investigational drug, etc.).
AUC[0-24]of rhTPO | For 9 days
  To assess plasma rhTPO Pharmacokinetic (PK) Parameter: Area under the concentration-time curve from time zero extrapolated to 24 hours(AUC [0-24]).
AUC [0-t] of rhTPO | For 9 days
  To assess plasma rhTPO PK Parameter: Area under the concentration-time curve from time zero to last time of quantifiable concentration(AUC [0-t]).
AUC [0-∞]of rhTPO | For 9 days
  To assess plasma rhTPO PK Parameter:
  area under the concentration-time curve from time zero extrapolated to infinity(AUC [0-∞]).
Cmax of rhTPO | For 9 days
  To assess plasma rhTPO PK Parameter：Observed maximum plasma concentration(Cmax).
tmax of rhTPO | For 9 days
  To assess plasma rhTPO PK Parameter：Time to Cmax (tmax).
t1/2 of rhTPO | For 9 days
  To assess plasma rhTPO PK Parameter：Elimination half-life (t1/2).
MRT for rhTPO | For 9 days
  To assess plasma rhTPO PK Parameter：Mean residence time (MRT).
Kel of rhTPO | For 9 days
  To assess plasma rhTPO PK Parameter：Elimination rate constant （Kel）.
Vd of rhTPO | For 9 days
  To assess plasma rhTPO PK Parameter：Apparent volume of distribution（Vd）.
CL/F of rhTPO | For 9 days
  To assess plasma rhTPO PK Parameter：apparent clearance (CL/F).

SECONDARY OUTCOMES:
Immunogenicity of rhTPO | Up to 12 months
  To evaluate the incidence of anti-rhTPO antibodies and neutralizing antibodies
Change of Platelet count (PLT) | Up to 29 days
  To evaluate the changing curve of platelet count (PLT) in each arm of subjects

CONTACTS AND LOCATIONS:
Locations (1):
- 302 Military Hospital of China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided